CLINICAL TRIAL: NCT04350229
Title: Endocrinological Changes Due to Pre-medications of Chemotherapy in Patients With Breast Cancer
Acronym: ALTEDEXAMAMA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto do Cancer do Estado de São Paulo (Other)
Responsible Party: Principal Investigator, Vanessa Armenio Scontre, Principal Investigator, Instituto do Cancer do Estado de São Paulo
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NP 1521/19
Record Dates: First submitted 2020-04-13; First posted 2020-04-16 (Actual); Last update posted 2023-10-05 (Actual); Status verified 2023-10

CONDITIONS: Breast Cancer
Keywords: breast cancer; endocrinological changes; dexamethasone
MeSH Terms: conditions — Breast Neoplasms | interventions — Control Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EXPERIMENTAL GROUP (Experimental): In the experimental group, dexamethasone will be omitted from the second application of paclitaxel.
  Pre-chemotherapy with the AC protocol: ondansetron 8mg and dexamethasone 10mg + Pre-chemotherapy with paclitaxel: ranitidine 50mg, ondansetron 8mg, diphenhydramine 50mg.
  Interventions: Drug: Drug omission
- CONTROL GROUP (Active Comparator): Pre-chemotherapy with the AC protocol: ondansetron 8mg and dexamethasone 10mg + Pre-chemotherapy with paclitaxel: ranitidine 50mg, ondansetron 8mg, diphenhydramine 50mg and dexamethasone 10mg.
  Interventions: Other: Control group

INTERVENTIONS:
Drug: Drug omission — Drug omission. In the experimental group, dexamethasone will be omitted from the second application of paclitaxel.
  Arms: EXPERIMENTAL GROUP
Other: Control group — No drug omission. In the control group, dexamethasone will not be omitted in the second application of paclitaxel.
  Arms: CONTROL GROUP

SUMMARY:
Treatment for patients with high-risk breast cancer diagnoses is based on chemotherapy drugs with side effects. Dexamethasone is a drug that is part of the arsenal of pre-chemotherapy medications to prevent adverse events resulting from treatment, however common endocrine pathological conditions resulting from high doses of this corticoid are clinically evident in these individuals. The aim of this study is to evaluate the omission of corticosteroid doses as a pre-medication in cancer treatment after the second week of treatment with taxane in a curative setting.

DETAILED DESCRIPTION:
Treatment for patients with diagnoses of high-risk breast cancer is based on chemotherapy drugs such as anthracyclines and taxanes and its main side effects described are cardiac toxicity and hypersensitivity and / or allergic reactions, respectively. Dexamethasone is a drug that is part of the arsenal of pre-chemotherapy medications to prevent adverse events resulting from treatment, however common endocrine pathological conditions resulting from high doses of this corticoid are clinically evident in these individuals.

These changes certainly have a negative impact on the patient's quality of life, however, with early recognition and the treatment of hypercortisolemia, we can lead to a reduction in morbidity and mortality in cancer patients.

The objective of this study is to evaluate whether the omission of corticosteroid doses as pre-medication in cancer treatment after the second week of treatment with taxane in a setting with curative intent can prevent or decrease the incidence of endocrinological changes, and what is its impact on treatment and on quality of life of the patient.

This is a prospective, randomized clinical study, without blinding as a research strategy used to increase the validity of clinical trials that evaluate the effect of interventions (eg, drugs or exercise). The process involves randomly assigning participants to an intervention group or to a control group and requires that participants have an equal chance of being allocated to either group.

Will be recruited 86 patients diagnosed with breast cancer with indication for neoadjuvant or adjuvant treatment with the standard ICESP protocol.

ELIGIBILITY:
Inclusion Criteria:

* Patients from the oncology services of ICESP and its Osasco unit.
* Over 18 years of age.
* Diagnosed with breast cancer who will be treated with an ACT Icesp scheme in the setting with curative intent (neoadjuvant and adjuvant).

Exclusion Criteria:

* Patients with significant cognitive impairment that prevents the questionnaire from being applied.
* Patients who are not fluent in Portuguese, or illiterate, who did not sign the ICF.
* ECOG 3 and KPS <70%.
* Metastatic patients, with the presence of other important morbidities that may interfere with laboratory findings.
* Patients with chronic use of steroidal and non-steroidal anti-inflammatory drugs.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2020-03-27 (Actual); Primary Completion 2022-06-20 (Actual); Study Completion 2022-06-20 (Actual)

PRIMARY OUTCOMES:
The incidence and change of endocrine dysfunction. | 36 months
  To evaluate the incidence and reduction of endocrine dysfunction in breast cancer patients with the administration of lower doses of dexamethasone in the solutions of pre-chemotherapy medications with doxorubicin, cyclophosphamide and paclitaxel (standard protocol AC-T of the ICESP).

SECONDARY OUTCOMES:
Inflammatory markers evaluation. | 36 months
  Evaluate inflammatory markers that may be related to endocrine syndromes resulting from the overuse of corticosteroids, and determine their correlation with the occurrence of endocrine syndromes.
Evaluation of the correlation between inflammatory markers and corticosteroid dose. | 36 months
  To assess the correlation between the serum level of inflammatory marker and the total dose of corticosteroids administered.
Progression Free Survival. | 36 months
  Progression-Free Survival (PFS) is defined as the time from registration to the earlier of progression or death due to any cause.
Change of Quality of life. | On the first day of treatment, on the first day of week 3 and on the last day of the final treatment.
  To compare change in Quality of Life, as defined by the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire Core-30 (EORTC QLQ-C30 (Version 3) during chemotherapy. The EORTC QLQ-C30 (Version 3) uses for the questions 1 to 28 a 4-point scale. The scale scores from 1 to 4: 1 ("Not at all"), 2 ("A little"), 3 ("Quite a bit") and 4 ("Very much"). Half points are not allowed. The range is 3.
  For the raw score, less points are considered to have a better outcome. The EORTC QLQ-C30 (Version 3) uses for the questions 29 and 30 a 7-points scale.
  The scale scores from 1 to 7: 1 ("very poor") to 7 ("excellent"). Half points are not allowed. The range is 6. First of all, raw score has to be calculated with mean values. Afterwards linear transformation is performed to be comparable. More points are considered to have a better outcome.
Cost change. | 36 months
  Analyze the treatment cost reduction omitting the use of dexamethasone in these patients.

CONTACTS AND LOCATIONS:
Overall Officials: Vanessa A Scontre, MD, Principal Investigator — Instituto do Cancer do Estado de São Paulo
Locations (1):
- Vanessa Scontre, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Undecided